CLINICAL TRIAL: NCT03829943
Title: Effects of Vitamin D on Human Sperm DNA Fragmentation
Brief Title: Vitamin D and Human Sperm DNA Fragmentation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanford Health (Other)
Responsible Party: Principal Investigator, Keith Hansen, Principal Investigator, Sanford Health
Other Study IDs: MOD00002311
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Infertility,Male; Vitamin D Deficiency
MeSH Terms: conditions — Infertility, Male; Vitamin D Deficiency | interventions — Vitamin D Response Element

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D deficiency: The study group will be males discovered to have Vitamin D deficiency.
  Interventions: Diagnostic Test: Vitamin D
- Control group: The control group will be males with normal Vitamin D status
  Interventions: Diagnostic Test: Vitamin D

INTERVENTIONS:
Diagnostic Test: Vitamin D — Blood will be drawn for Vitamin D level

SUMMARY:
The purpose of this study will be to investigate if there is a correlation between Vitamin D levels and Sperm DNA Fragmentation. This is a prospective, cohort study. In this study male participants presenting with their partners because of inability to conceive will be recruited for this study. Participants will have a blood sample drawn which will be tested for Vitamin D level. The investigators will then compare sperm DNA fragmentation between normal Vitamin D levels, Vitamin D insufficiency, and Vitamin D deficiency. All infertile males who present to the investigators' infertility clinic have a Semen analysis and Sperm chromatin Structure Assay (SCSA). The research part of the study will be to obtain the Vitamin D level.

DETAILED DESCRIPTION:
Vitamin D plays an important role in bone metabolism and has also been discovered to influence male reproduction. Vitamin D binds to the Vitamin D receptor which then can bind to Vitamin D response elements in the DNA which can alter transcription. By changing transcription it can have long term effects on cellular metabolism. Previous studies have demonstrated abnormalities in sperm motility and morphology in males who are Vitamin D deficient. The mechanism by which Vitamin D affects spermatogenesis (formation of sperm) is unknown. One possibly mechanism by which deficient Vitamin D may affect sperm formation is through DNA fragmentation. The head of the sperm contains all the DNA. When a sperm cell is made the DNA in the nucleus must be super compacted to accomplish sperm formation. To sufficiently compact the DNA, first the DNA is 'turned off' and then very tightly wound (or compacted) into toroids (like small tires) which are stacked one on top of another. During this process of compaction the DNA will occasionally break or fragment. The egg can repair the DNA fragmentation as long as there is not a large amount of breakage. If the DNA fragmentation exceeds a certain amount then fertilization and early development of the embryo may be adversely affected. DNA fragmentation can be tested by using the Sperm Chromatin Structure Assay (SCSA), which the investigators currently measure in males who present with their partners with infertility. Previous studies have suggested that the abnormalities in sperm due to vitamin D deficiency may be related to increased DNA fragmentation. This study will assist in understanding the cause of sperm abnormalities in subjects with Vitamin D deficiency.

This is a prospective, cohort study. In this study male patients who present with inability to conceive will be asked to be involved in this study. After agreement with the study, a blood sample drawn which will be tested for Vitamin D level. The investigators will then compare sperm DNA fragmentation between normal Vitamin D levels, Vitamin D insufficiency, and Vitamin D deficiency. All infertile males presenting to the investigators' infertility clinic have a Semen analysis and Sperm chromatin Structure Assay (SCSA). The research part of the study will be to obtain the Vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* Male with diagnosis of infertility.

Exclusion Criteria:

* Azoospermia

Ages: 21 Years to 56 Years | Sex: Male
Age Groups: Adult
Study Population: Male partners of infertile couples. All males who present to our Infertility clinic will be offered participation.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Sperm DNA Fragmentation | 1 year
  Human Sperm DNA fragmentation will be determined by the Sperm Chromatin Structure Assay.

SECONDARY OUTCOMES:
High DNA stainability | 1 year
  High DNA stainability is determined by the Sperm Chromatin Structure Assay and is consistent with immature sperm.
Sperm density | 1 year
  This will be determined by microscopic analysis of participant's semen and expressed as millions per milliliter

OTHER OUTCOMES:
Sperm motility | 1 year
  This will be determined by microscopic analysis of participant's semen and expressed as percent motile.
Sperm morphology | 1 year
  This will be determined by microscopic analysis of participant's semen and will be expressed as percent normal forms.
Height | 1 year
  Measured by stadiometer and recorded in centimeters.
Weight | 1 year
  Measured using digital, medical scale
BMI | 1 year
  weight and height will be combined to report BMI in kg/m^2
Tobacco status | 1 year
  Patient will be asked if uses tobacco products: smoke, smokeless
Race/ethnicity | 1 year
  Patient will self identify race/ethnicity

CONTACTS AND LOCATIONS:
Locations (1):
- Sanford Health Fertility and Reproductive Medicine, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share individual participant data (IPD) with researchers who desire information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after collection complete and will remain available for 3 years.
Access Criteria: Investigator.

REFERENCES:
- [Background] Blomberg Jensen M, Bjerrum PJ, Jessen TE, Nielsen JE, Joensen UN, Olesen IA, Petersen JH, Juul A, Dissing S, Jorgensen N. Vitamin D is positively associated with sperm motility and increases intracellular calcium in human spermatozoa. Hum Reprod. 2011 Jun;26(6):1307-17. doi: 10.1093/humrep/der059. Epub 2011 Mar 22. PMID 21427118
- [Background] Bunde E, Hanssen K, Huntington MK. Vitamin D status in eastern South Dakota. S D Med. 2012 Jun;65(6):227, 229, 231. PMID 22856011
- [Background] Boisen IM, Bollehuus Hansen L, Mortensen LJ, Lanske B, Juul A, Blomberg Jensen M. Possible influence of vitamin D on male reproduction. J Steroid Biochem Mol Biol. 2017 Oct;173:215-222. doi: 10.1016/j.jsbmb.2016.09.023. Epub 2016 Sep 28. PMID 27693423
- [Background] Blomberg Jensen M, Lawaetz JG, Petersen JH, Juul A, Jorgensen N. Effects of Vitamin D Supplementation on Semen Quality, Reproductive Hormones, and Live Birth Rate: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Mar 1;103(3):870-881. doi: 10.1210/jc.2017-01656. PMID 29126319
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM. Guidelines for preventing and treating vitamin D deficiency and insufficiency revisited. J Clin Endocrinol Metab. 2012 Apr;97(4):1153-8. doi: 10.1210/jc.2011-2601. Epub 2012 Mar 22. No abstract available. PMID 22442274